CLINICAL TRIAL: NCT03446326
Title: Assessment of Stroke Volume and Cardiac Output in Response to Varying Heart Rates and Body Position - a Pacemaker Based Study
Brief Title: Assessment of Stroke Volume and Cardiac Output in Response to Varying Heart Rates
Acronym: Pacing_SV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB15-2887
Record Dates: First submitted 2018-01-31; First posted 2018-02-26 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Vasovagal Syncope
Keywords: pacemaker; stroke volume; cardiac output; heart rate
MeSH Terms: conditions — Syncope, Vasovagal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Stroke volume and cardiac output (Experimental): Pacing runs will occur at the following rates:
  * 50 beats per minute (bpm)
  * 60 bpm
  * 70 bpm
  * 80 bpm
  * 90 bpm
  * 100 bpm
  * 110 bpm
  * 120 bpm
  * 130 bpm
  The finger blood pressure cuff will be calibrated between pacing runs.
  Following the final pacing run while supine, the patient will be given 10 minutes to rest prior to the upright portion of the study. They will then be strapped into the table (so they will not fall) and then they will be tilted up to >70 degrees (almost standing up). They will stand for ~10 minutes prior to commencing the next pacing trains.
  Interventions: Device: Pacing

INTERVENTIONS:
Device: Pacing — Assess the non-invasively determined stroke volume and cardiac output response at different paced heart rates in patients with a cardiac pacemaker or implanted defibrillator with preserved ejection fractions (LVEF≥50%)

SUMMARY:
The investigators will seek to determine the effects of different heart rates on both stroke volume and cardiac output using non-invasive hemodynamic assessments. In order to safely manipulate the HR, the investigators will study patients with permanent pacemakers in whom heart rate manipulation can be done in a safe and non-invasive manner.

DETAILED DESCRIPTION:
Permanent pacemakers have sometimes been used to treat patients with recurrent vasovagal syncope. This is because patients with vasovagal syncope often experience bradycardia at the time of their syncope. Unfortunately, pacemakers are often ineffective in preventing syncope.

Classical cardiovascular hemodynamics would suggest that increasing the heart rate (HR; via pacemaker) should increase the cardiac output (CO). This is because:

CO = HR x Stroke volume (SV).

The assumption is that the SV is fixed during manipulation of the HR. However, this might not be the case. As the number of beats per minute (HR) increases, the cardiac cycle length (R-R interval [RRI]) shortens, as a function of simple math. This means that the time in cardiac systole shortens, and the time in cardiac diastole shortens. Since cardiac diastole is when the heart fills up with blood, faster HR can be associated with decreased cardiac filling times. This, in turn, could compromise the SV. However, there is a paucity of data as to what happens to SV and CO at different HR. Further, it is possible that these effects will be different when a person is lying down supine versus when a patient is upright (when stroke volume will be lower).

The investigators will seek to determine the effects of different HR on both SV & CO. In order to safely manipulate the HR, they will study patients with permanent pacemakers in whom HR manipulation can be done in a safe and non-invasive manner.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years (inclusive)
* Implanted permanent pacemaker or implanted defibrillator capable of atrial and ventricular pacing
* LV ejection fraction >50%

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Clinical need for a cardiac resynchronization device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac output while atrial pacing at lower and higher rates while supine | 1 day
  Change in cardiac output (CO) when atrial pacing at 80 bpm & 120 bpm while supine. CO = HR x Stroke volume (SV)

SECONDARY OUTCOMES:
Change in cardiac output at lower and higher ventricular (VVI) paced rates while supine | 1 day
  Change in Cardiac output at ventricular (VVI) paced rates when it is lower (50-70 bpm) and higher (130 bpm) while supine
Change of cardiac output at lower and higher atrial (AAI) paced rates while supine versus while upright | 1 day
  Change of cardiac output at lower and higher atrial (AAI) paced rates while supine versus while upright at different paced rates
Change of cardiac output at lower and higher ventricular (VVI) paced rates while supine versus while upright | 1 day
  Change of cardiac output at lower and higher ventricular (VVI) paced rates while supine versus while upright at different paced rates
Change in stroke volume at lower and higher atrial paced rates while tilted up | 1 day
  Change in stroke volume at lower (50-70 bpm) vs. higher (130 bpm) atrial paced rates while tilted up
Change in stroke volume at lower and higher ventricular (VVI) paced rates while tilted up | 1 day
  Change in stroke volume at ventricular (VVI) paced rates when it is lower (50-70 bpm) and higher (130 bpm) while tilted up
Change of stroke volume at lower and higher atrial (AAI) paced rates while supine versus while upright | 1 day
  Change of stroke volume at lower and higher atrial (AAI) paced rates while supine versus while upright at different paced rates
Change of stroke volume at lower and higher ventricular (VVI) paced rates while supine versus while upright | 1 day
  Change of stroke volume at lower and higher ventricular (VVI) paced rates while supine versus while upright at different paced rates

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No